CLINICAL TRIAL: NCT05582382
Title: Validation of Prognostic Clinical Risk Scores in Predicting Outcomes for Patients Diagnosed With COVID-19 During Initial Triage Assessment
Brief Title: Validation of Prognostic Clinical Risk Scores in Predicting Outcome for Patients With COVID-19 at Initial Triage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr Adnan Agha (Other)
Collaborators: Abu Dhabi Health Services Company (Other Government)
Responsible Party: Sponsor-Investigator, Dr Adnan Agha, Assistant Professor, Internal Medicine, College of Medicine and Health Sciences, United Arab Emirates University, United Arab Emirates University
Organization: United Arab Emirates University (Other)
Other Study IDs: CMHS_IntMed_DOH/CVDC/2020/1251
Record Dates: First submitted 2022-10-14; First posted 2022-10-17 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: hospitalization; COVID-19; clinical risk score; morbidity; prediction
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: logistic regression of known prognostic markers of severity of COVID19 — An observational longitudinal follow up of all consecutive patients with positive SARS-CoV-2 testing on nasopharyngeal swabs per WHO definitions presenting to the emergency department . The risk assessment score at initial presentation will be calculated for each patient using clinical assessment scoring of ALA & ALKA and compared with the currently proposed clinical risk assessment scoring system
  The utility of the risk score in triaging patients on their initial visits to emergency department (ED) will be validated against the following measured outcomes:
  1. Hospital admission on the first encounter to ED
  2. Admission to ICU for the duration of the COVID-19 hospitalization
  3. In hospital and out of hospital mortality
  4. Return to ED following initial discharge (within the current covid illness period, Maximum 30 days from the initial diagnosis)

SUMMARY:
Background Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) causing Covid-19 pandemic continues to be a global health threat with a massive burden on health care systems resulting in more than six million deaths in 188 countries. Because of wide clinical spectrum of disease severity, having clinically applicable prognostic tools for early identification of patients at high risk of progression to severe / critical illness is essential to guide clinical decision making and resource allocation efforts. So far, clinical prognostic tools have focused on host factors, but more recent data indicated a significant association between SARS-CoV-2 variants and the development of complications such as long COVID.

Objectives

1. Validation of the ALA & ALKA prediction tools for initial evaluation of patients diagnosed with COVID-19 infection.
2. Comparison of performance of the ALA & ALKA prediction tools with the currently clinical risk assessment scoring system used during initial evaluation of patients diagnosed with COVID-19 infection.
3. Evaluation of the clinical risk assessment scoring based on number of comorbidities in prediction of COVID-19 related complications
4. Assessment of the association between SARS-CoV-2 variants and the risk of COVID-19 severity
5. Assessment of the impact of SARS-CoV-2 variants on the performance of ALA & ALKA prediction tools

Methods Data will be abstracted from electronic medical records including demographics, clinical manifestation, comorbidities, and initial laboratory data in patients with Covid 19 infection of around 2000 patients presented initially to COVID assessment centre, including SARS CoV-2 sequencing data. Furthermore, population level SARS-CoV-2 RNA sequence data will also be examined and correlated with COVID-19 severity and the performance of prediction tools.

DETAILED DESCRIPTION:
Background:

Since December 2019, when severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) causing COVID -19 disease emerged in Wuhan city and on 11 March 2020 rapidly spread into the rest of the world including UAE as a pandemic. COVID-19 continues to be a global health threat with a massive burden on health care systems resulting in more than six million deaths in 188 countries (1).

COVID-19 infection is characterized by a wide clinical spectrum of disease severity ranging from asymptomatic illness to severe disease that may progress to life-threatening complications such as shock and acute respiratory distress syndrome (2). Thus, having clinically applicable prognostic tools for early identification of symptomatic patients at high risk of progression to severe / critical illness is essential to guide allocating limited healthcare resources (3). So far, clinical prognostic tools have focused on host factors, but more recent data indicated a significant association between SARS-CoV-2 variants and the development of complications such as long COVID (4).

Currently, the clinical assessment for patients with COVID-19 infection is based on patient's age, number of comorbidities, subjective symptoms, and extent of pulmonary infiltrate on radiological examination which makes early prediction of severe / critical illness rather difficult (5-7). A recently published prognostic prediction tools (ALA & ALKA) were proposed to aid triaging patients with COVID-19 infection on initial diagnosis (8). These prediction tools are based on simple readily available laboratory tests and therefore may offer a clear advantage over other tools to guide discharge and admission decisions in triage assessment centers Nevertheless, external validation of these simple tools using another cohort of patients would provide a stronger evidence to support their utility in triaging patients on initial diagnosis. In addition, it will also allow further optimization of these tools to improve their utility as clinical decision support tools to triage patients on initial diagnosis. Patients deemed to be high risk based on these predictive tools could be triaged to hospital admission where intensive care unit (ICU) is available in anticipation of worse outcome. Therefore, these patients may benefit from earlier initiation of the required level of care and support including specific therapy.

The aim of this study is to validate and compare the ALA & ALKA prediction tools with the currently clinical risk assessment scoring system proposed for initial evaluation of patients with COVID-19 infection.

Methodology:

An observational longitudinal follow up of all consecutive patients with positive SARS-CoV-2 testing on nasopharyngeal swabs per WHO definitions presenting to the emergency department . Furthermore, population level SARS-CoV-2 RNA sequence data will also be examined and correlated with COVID-19 severity and the performance of prediction tools.

Data will be abstracted from electronic medical records using a data collection tool. This includes demographics, clinical manifestation, number of comorbidities, initial laboratory and radiological examination results and their final outcomes as detailed below.

The risk assessment score at initial presentation will be calculated for each patient using clinical assessment scoring of ALA & ALKA and compared with the currently proposed clinical risk assessment scoring system

The utility of the risk score in triaging patients on their initial visits to emergency department (ED) will be validated against the following measured outcomes:

1. Hospital admission on the first encounter to ED
2. Admission to ICU for the duration of the COVID-19 hospitalization
3. In hospital and out of hospital mortality
4. Return to ED following initial discharge (within the current covid illness period, Maximum 30 days from the initial diagnosis)

Sample Collection Process:

Data will be abstracted from electronic medical records using a data collection tool. The data would include demographics, clinical manifestation, comorbidities, laboratory and radiological results, and final outcomes.

The assessment risk score at initial presentation will be calculated using a free web-based online calculator.

Data Handling & Analysis:

Descriptive statistics will be generated for all variables. Multivariate logistic regression models to fit for outcomes. Variables incorporated in the COVID-19 risk of score will be included in the regression analysis to predict the outcomes. Multivariate logistic regression results will be presented in terms of adjusted Odds Ratios with corresponding 95% confidence intervals and p-values.

Discrimination will be evaluated using C-Statistic, along with its corresponding 95% Confidence Intervals and Receiver Operating Characteristic (ROC) curve. C-Statistics ≥ 0.7 will be considered good and ≥ 0.8 will be considered excellent (9). Calibration will be assessed based on the predicted probability for the outcome as predicted from the regressions. Calibration curves will be generated. P-values <0.05 is considered statistically significant. All analysis will be performed using SPSS software (version 28, IBM Corp, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with positive SARS-CoV-2 testing on nasopharyngeal swabs per WHO definitions presenting to the emergency department
* All patients admitted to the hospital for isolation purposes only

Exclusion Criteria:

* Inconclusive PCR results on initial or repeat results with 24 hours

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The sample will include all consecutive symptomatic patients with confirmed COVID-19 infection presented to ED. A sample size of 2000 is required for the validation of the prognostic predictive tools.
  Sample Collection Process:
  Data will be abstracted from electronic medical records using a data collection tool. The data would include demographics, clinical manifestation, comorbidities, laboratory and radiological results, and final outcomes.
  The assessment risk score at initial presentation will be calculated using a free web-based online calculator.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Validation of the ALA & ALKA prediction tools | 12 months
  Validation of the ALA & ALKA prediction tools for initial evaluation of patients diagnosed with COVID-19 infection

SECONDARY OUTCOMES:
Comparison of performance of the ALA & ALKA prediction tools with current clinical risk tools | 12 months
  Comparison of performance of the ALA & ALKA prediction tools with the currently clinical risk assessment scoring system used during initial evaluation of patients diagnosed with COVID-19 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Agha, Principal Investigator — United Arab Emirates University
Locations (1):
- Internal Medicine, College of Medicine and Health Sciences, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
Non identifiable data for this validation study upon completion will be released for researchers including performance of individual markers of severity as well as final model

REFERENCES:
- [Background] Wiersinga WJ, Rhodes A, Cheng AC, Peacock SJ, Prescott HC. Pathophysiology, Transmission, Diagnosis, and Treatment of Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 Aug 25;324(8):782-793. doi: 10.1001/jama.2020.12839. PMID 32648899
- [Background] Halalau A, Imam Z, Karabon P, Mankuzhy N, Shaheen A, Tu J, Carpenter C. External validation of a clinical risk score to predict hospital admission and in-hospital mortality in COVID-19 patients. Ann Med. 2021 Dec;53(1):78-86. doi: 10.1080/07853890.2020.1828616. Epub 2020 Oct 9. PMID 32997542
- [Background] Dardenne N, Locquet M, Diep AN, Gilbert A, Delrez S, Beaudart C, Brabant C, Ghuysen A, Donneau AF, Bruyere O. Clinical prediction models for diagnosis of COVID-19 among adult patients: a validation and agreement study. BMC Infect Dis. 2022 May 14;22(1):464. doi: 10.1186/s12879-022-07420-4. PMID 35568825
- [Background] Kurban LAS, AlDhaheri S, Elkkari A, Khashkhusha R, AlEissaee S, AlZaabi A, Ismail M, Bakoush O. Predicting Severe Disease and Critical Illness on Initial Diagnosis of COVID-19: Simple Triage Tools. Front Med (Lausanne). 2022 Feb 10;9:817549. doi: 10.3389/fmed.2022.817549. eCollection 2022. PMID 35223916